CLINICAL TRIAL: NCT00958178
Title: A Novel Method of Preoxygenation Using Partial Rebreathing Via a Coaxial Mapleson D Breathing System (Bain Circuit)
Brief Title: A Novel Method of Preoxygenation Using a Bain Circuit
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: John Glen, National Health Service
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08/S071038
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rebreathing method of preoxygenation (Experimental): Subjects will breathe Oxygen through a close fitting mask, but the flow will be low so that they rebreathe some of their expired air. After 30 seconds, the flow will be turned up so that they will breathe 100% Oxygen.
  Interventions: Drug: Oxygen
- T method of preoxygenation (Active Comparator): Tidal breathing of 100% oxygen through a well fitting facemask, for 4 minutes.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Experimental: Low flow Oxygen for 30 seconds then high flow for 3.5 minutes. Active comparator: High flow Oxygen for 4 minutes.

SUMMARY:
The purpose of this study is to determine whether rebreathing for a short time (a bit like breathing into a paper bag) will stimulate faster breathing and thus make the giving of Oxygen more effective.

The hypothesis is that the investigators method (rebreathing) will be faster than the current method of administering Oxygen.

DETAILED DESCRIPTION:
It is standard practice for patients to breathe oxygen before receiving a general anaesthetic. This is called preoxygenation. It is done by using a mask which fits snugly onto the face. But for how long should patients breathe oxygen? Is taking deep breaths a good idea? What is the best oxygen flow rate? These questions are important because preoxygenation is one of the things which makes anaesthesia safe, so finding the best way of doing it might help save lives. Previous research has attempted to identify the best way to give oxygen before anaesthesia. It seems that breathing pure oxygen for three minutes is enough, or if you are in an urgent situation, then taking deep breaths of pure oxygen for a minute will do. However, there is another possible way of doing it which has not yet been looked at.

Asking someone to breathe back in the air they have just exhaled seems, on the face of it, to be pointless at best. But doing just that for a very short time will make the person breathe harder. Then when you give them pure oxygen, they will breathe it in really deeply and this might make the preoxygenation quicker. That's the theory. To test it we plan to ask 40 healthy people to do the standard preoxygenation, then try our new way. We won't be giving anaesthetic, just the oxygen.

The hypothesis is that our new method will be quicker than the existing one.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-27
* Non-smoker
* No chronic cardiorespiratory or neuromuscular illness
* No intercurrent illness

Exclusion Criteria:

* Unable/unwilling to consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Time to end-tidal oxygen of 90% | 5 minutes

SECONDARY OUTCOMES:
Level of discomfort as assessed by questionnaire | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: John Glen, MBChB, Principal Investigator — UK National Health Service
Locations (1):
- Victoria Infirmary, Glasgow, Glasgow, United Kingdom